CLINICAL TRIAL: NCT07145515
Title: Enhancing Heart Allograft Function With the OCS Heart System (ENHANCE) Trial
Brief Title: Enhancing Heart Allograft Function With the OCS Heart System Trial
Acronym: ENHANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCS-HEART-031725
Record Dates: First submitted 2025-08-25; First posted 2025-08-28 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Heart Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Part A (OCS Heart) (Experimental): DCD Donor Hearts & DBD Donor Hearts Initially Deemed Unsuitable for Cold Storage (Current Approved Indications)
  Interventions: Device: OCS Heart
- Part B (OCS Heart) (Experimental): DBD Donor Hearts Currently Used with Cold Storage
  Interventions: Device: OCS Heart
- Part B (SCS) (Active Comparator): DBD Donor Hearts Currently Used with Cold Storage
  Interventions: Other: Static Cold Storage (SCS)

INTERVENTIONS:
Device: OCS Heart — Preservation of donor hearts with OCS Heart System and novel OCS Solution and OCS Functional Enhancer.
  Arms: Part A (OCS Heart); Part B (OCS Heart)
Other: Static Cold Storage (SCS) — Preservation of donor hearts with static cold storage.
  Arms: Part B (SCS)

SUMMARY:
This trial is designed to evaluate the safety and effectiveness of the novel OCS Solution and OCS Functional Enhancer (OFE) to support FDA approval in both DBD and DCD heart transplantation. In addition, this trial will evaluate the performance of the novel OCS Solution and OFE compared to Static Cold Storage (SCS) in DBD heart transplantation to potentially demonstrate superiority.

ELIGIBILITY:
Part A - DCD Donor Hearts & DBD Donor Hearts Initially Deemed Unsuitable for Cold Storage (Current Approved Indications):

Donor Inclusion Criteria

* Donor hearts are deemed clinically acceptable for transplantation after physical examination of the donor hearts in the donor chest and/or on the back table in the donor operating room.
* All DCD donors eligible for functional warm ischemic time criteria ≤ 30 minutes. WIT defined as time from when mean systolic blood pressure (SBP) is <50mmHg (sustained for at least 5 minutes) to aortic cross clamp and administration of old cardioplegia in the donor.
* DBD donor hearts with an expected cross clamp of ≥ 4 hours
* DBD donor hearts with any of the following organ quality concerns, regardless of cross clamp time:

  * Donor age ≥ 40 years old
  * Unknown downtime
  * Insignificant CAD
  * LVEF ≤ 50%

Donor Exclusion • Moderate to severe aortic incompetence

Part B - DBD Donor Hearts Currently Used with Cold Storage (New Indication):

Donor Inclusion Criteria

* Donor hearts are deemed clinically acceptable for transplantation after physical examination of the donor hearts in the donor chest and/or on the back table in the donor operating room.
* Eligible for randomization to OCS or SCS treatment arms.
* DBD donor hearts with an expected cross clamp time of < 4 hours.

Donor Exclusion

* Moderate to severe aortic incompetence
* DBD donor with any of the following organ quality concerns:

  * Donor age ≥ 40 years old
  * Unknown downtime
  * Insignificant CAD
  * LVEF ≤ 50%

Recipient Eligibility Criteria (for Part A and B Cohorts)

Inclusion

* Signed informed consent document and authorization to use and disclose protected health information
* Heart transplant candidate
* Age ≥ 18 years old

Exclusion

• Participant in any other interventional clinical or investigational trials/programs that may confound the outcomes of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Patient and graft survival | 30-day post transplant
  The primary endpoint is 30-day patient and graft survival with freedom from moderate or severe LV or RV primary graft dysfunction (PGD) in the first 24 hours post-transplant.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California San Francisco, San Francisco, California
  - Tampa General Hospital, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mount Sinai, New York, New York
  - Columbia University Irving Medical Center/ New York Presbyterian Hospital, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Duke University, Durham, North Carolina
  - Baylor Scott and White, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No